CLINICAL TRIAL: NCT04817345
Title: Peripheral Blood Stem Cell Collection From Patients With Sickle Cell Disease (SCD) Using Plerixafor
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The safety and efficacy of plerixafor in adult and pediatric SCD patients was an unknown when we started. A lot more data from therapeutic trials is available. We feel that recruiting patients without a therapeutic option isn't ethically justifiable.
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: Doris Duke Charitable Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: ASPIRES2
Record Dates: First submitted 2021-03-23; First posted 2021-03-26 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Sickle Cell Disease
Keywords: Plerixafor; Leukapheresis; Mobilization; Stem Cells; Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — plerixafor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Plerixafor (Experimental): Participants will receive a subcutaneous dose of 0.24 mg/kg of plerixafor once daily (Q24hr) x 2 days.
  Interventions: Drug: Plerixafor

INTERVENTIONS:
Drug: Plerixafor — Subcutaneous
  Other Names: Mozobil ™

SUMMARY:
With recent advances in gene editing, gene therapy is becoming a viable curative treatment option for sickle cell disease. In order to do genetic manipulation, investigators need to collect hematopoietic stem cells from patients with sickle cell disease. In this study, investigators want to study the safety and feasibility of collecting peripheral blood stem cells from pediatric and young adult patients with sickle cell disease after administering plerixafor. Studying these peripheral blood stem cells will help in optimizing the yield of peripheral CD34+ cells from pediatric and young adult patients with sickle cell disease, which in turn will help to develop better gene therapies for these patients.

Primary Objectives

* Determine the safety profile associated with administration of plerixafor in pediatric and young adult patients with sickle cell disease (SCD).
* To estimate the number of CD34+ cells/kg of body weight that can be collected with peripheral apheresis after administration of plerixafor in pediatric and young adult patients with SCD.

Exploratory Objectives

* To describe the kinetics of CD34+ cell mobilization in peripheral blood after - + cells obtained from pediatric and young adult patients with SCD.
* To study the effect of hydroxyurea therapy on senescence in plerixafor-mobilized CD34+ cells obtained from pediatric and young adult patients with SCD.

DETAILED DESCRIPTION:
Participants will be enrolled sequentially, and no two participants will undergo drug administration, mobilization or apheresis at the same time. A subsequent participant can only receive the study drug when the previous participant has been safely apheresed and discharged from the hospital. In the first stratum of the study only adult participants (18-25 years of age) will be enrolled. Once plerixafor and apheresis has been shown to be safe and acceptable in at least 5 adult participants, the study will enroll participants in the pediatric stratum. Pediatric stratum will not be activated until all the patients in the adult stratum have been evaluated and completed participation with acceptable results. In the pediatric stratum, older children (14 years old and above) will be enrolled before younger children (10-14 years old). After 10 participants, 14 years and older, have safely completed the study participation, younger children 10-14 years old will be allowed to participate.

Prophylactic red blood cell exchange or simple red cell transfusions will be given within 7 days prior to plerixafor administration to participants targeting HbS <30% to reduce the incidence of vaso-occlusive crisis and other events that may be associated with high hemoglobin S levels.Hydroxyurea treatment should be stopped 4 weeks before mobilization. Plerixafor administration and apheresis will be timed for participants already receiving chronic transfusion therapy such that the plerixafor administration and apheresis coincides with regularly timed transfusion.

Participants undergoing hematopoietic stem cell (HSC) mobilization will receive a daily-dose subcutaneous administration of plerixafor (Mozobil®) at 0.24 mg/kg on up to 2 consecutive days. Leukapheresis will start approximately 4 hours after each dose of plerixafor is given. This process lasts 4-10 hours.

Participants will be followed for 30 days after the last dose of plerixafor and then taken off study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with severe SCD who are 10-25 years old and are willing to donate autologous HSCs for advancing future gene therapy for SCD. Parents/legal guardians of participants must be able and willing to consent for their participation in this study. Severe SCD, for the purpose of this study, will be defined as patients who are receiving chronic transfusion therapy due to SCD related complications. The need for undergoing chronic transfusion therapy must be determined by the primary hematologist. Some patients may continue to receive hydroxyurea in addition to and simultaneously with blood transfusion therapy. Such patients are eligible for inclusion on the study if they hold hydroxyurea for at least 4 weeks. The ability to hold hydroxyurea (or not) with ongoing chronic transfusion therapy will be made by the primary hematologist as well. All genotypes of SCD will be eligible.
* Adequate renal function: serum/plasma creatinine < 1.5 mg/dL and creatinine clearance > 50 mL/min (as calculated by the Crockcroft-Gault formula).
* Adequate liver function: direct bilirubin < 2.5 times the upper limit of normal range, AST and ALT < 5 times the upper limit of normal range.
* Blood counts: WBC > 3,000/mm^3, granulocytes > 1,000/mm^3, hemoglobin > 7.0 g/dL, platelets > 150,000/mm^3.
* Female patients of childbearing age should have a negative serum pregnancy test within one week of beginning plerixafor administration, have had a hysterectomy, be post-menopausal.
* Negative serologic tests for syphilis, hepatitis B and C, HIV, and HTLV-1/II.
* Participants should either have a central line in place or be able to undergo apheresis without the necessity of the insertion of a central venous catheter
* Participants of childbearing potential should agree to use of an effective form of contraception during treatment and for at least 1 week after the last dose of plerixafor.
* ECOG performance status/Karnofsky score/Lansky score >80.

Exclusion Criteria:

* Pregnancy. Female patients of childbearing age should have a negative serum pregnancy test within one week of beginning plerixafor administration, except those that have had a hysterectomy, or are post-menopausal.
* Active viral, bacterial, fungal, or parasitic infection.
* History of cancer, excluding squamous carcinoma of the skin and cervical carcinoma in situ.
* Active and painful splenomegaly or splenomegaly (size greater than upper limit of normal) or splenic sequestration determined by ultrasound.
* Previous history of splenomegaly or splenic sequestration, unless HbS level of <30% is documented within 48-72 hours of each plerixafor dose
* Allergy to plerixafor.
* Patients receiving hydroxyurea will not be included in the study. However, they may be included if the primary hematologist determines that hydroxyurea can be safely discontinued for at least 4 weeks prior to the plerixafor administration and apheresis. Generally, patients receiving chronic transfusion therapy can safely discontinue hydroxyurea therapy as there is unlikely to be any added benefit, but this will be determined by the primary treating hematologist.
* Poor cardiac function, as defined by an ejection fraction < 40%.
* History of clinically proven pulmonary hypertension.
* Emergency room admission or hospitalization in the past 14 days prior to first dose of study drug.
* Major surgery in the past 30 days prior to first dose of study drug.

Ages: 10 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2023-04 (Estimated); Primary Completion 2023-04 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Number of participants with sufficient collection of hematopoietic stem cells (HSCs) without serious adverse events. | 2 days
  Sufficient collection of HSCs from peripheral blood after plerixafor mobilization without serious adverse events (SAEs)

CONTACTS AND LOCATIONS:
Overall Officials: Akshay Sharma, MBBS, Principal Investigator — St. Jude Children's Research Hospital; Mitch Weiss, MD, PhD, Principal Investigator — St. Jude Children's Research Hospital

IPD SHARING:
Plan to Share IPD: Yes
Individual participant de-identified datasets containing the variables analyzed in the published article will be made available (related to the study primary or secondary objectives contained in the publication). Supporting documents such as the protocol, statistical analyses plan, and informed consent are available through the CTG website for the specific study. Data used to generate the published article will be made available at the time of article publication. Investigators who seek access to individual level de-identified data will contact the computing team in the Department of Biostatistics (ClinTrialDataRequest@stjude.org) who will respond to the data request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available at the time of article publication.
Access Criteria: Data will be provided to researchers following a formal request with the following information: full name of requestor, affiliation, data set requested, and timing of when data is needed. As an informational point, the lead statistician and study principal investigator will be informed that primary results datasets have been requested.

REFERENCES:
- See also: St. Jude Children's Research Hospital — https://www.stjude.org
- See also: Clinical Trials Open at St. Jude — https://www.stjude.org/protocols